CLINICAL TRIAL: NCT03002896
Title: A Pilot Study of a Mobilized Psychoeducation and Skills Based Intervention (Pep-Pal) for Caregivers of Patients With Advanced Illness
Brief Title: Mobilized Psychoeducation and Skills Based Intervention (Pep-Pal) for Caregivers of Patients With Advanced Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16-0990
Record Dates: First submitted 2016-09-28; First posted 2016-12-26 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Distress; Anxiety; Depression
Keywords: Cancer; Caregivers; Pep-pal; Pep-Pal + Treatment as Usual; Treatment as Usual
MeSH Terms: conditions — Anxiety Disorders; Depression; Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pep-Pal + Treatment as Usual (Experimental): If the caregiver is assigned to the Pep-Pal intervention condition, the RA will provide access to the mobilized website (passcode) through an email. Caregivers will be instructed to watch each session at least once. It will be recommended that caregivers watch one to two new sessions per week so that they can have enough time to practice the skills between sessions. In addition, they will be told that they can go back and watch the sessions for review as many times as they like. Full participation will be defined as watching at least 7/9 sessions (75% of program) based on previous criteria for similar intervention completion in a prior trial with advanced cancer patients.
  Interventions: Behavioral: Pep-Pal; Other: Treatment as Usual
- Treatment as Usual (Active Comparator): Treatment as usual provides voluntary (at the caregiver's discretion) support services for the caregivers which is rarely used by the caregivers.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Pep-Pal — Pep-Pal is designed to complement the utilization of other resources, provide support when no other resources can be obtained, or provide support in the interim until greater resources can be obtained. In this way, Pep-Pal is a resource for our most hard to reach caregivers.
  Arms: Pep-Pal + Treatment as Usual
Other: Treatment as Usual

SUMMARY:
The proposed project is a pilot study of the Pep-Pal (Psychoeducation and Skills Based Intervention) versus a treatment as usual control group. A total of 60 caregivers; including caregivers of patients with HSCT (Hematopoietic Stem Cell Transplantation), caregivers enrolled in Phase I clinical trials, and caregivers of patients with advanced cancer (Stage III, solid tumor) will be enrolled in this study. The investigators do not expect different outcomes from these three groups, rather these populations are selected to optimize recruitment within a short time frame. The caregivers will be randomized to either treatment as usual or Pep-Pal intervention.

DETAILED DESCRIPTION:
The proposed project is a pilot study of the Pep-Pal intervention versus a treatment as usual control group. A total of 60 caregivers; caregivers of patients with HSCT, caregivers of patients enrolled in phase I oncology trials, and caregivers of patients with advanced cancer (Stage IV, solid tumor) will be enrolled in this study. The investigators do not expect different outcomes from these three groups, rather these populations are selected to optimize recruitment within a short time frame. The caregivers will be randomized to either treatment as usual or Pep-Pal intervention. The proposed study population is based on prior research indicating that caregivers of patients receiving HSCT, caregivers of patients enrolled in phase I oncology trials, and caregivers of patients with advanced cancer experience significant distress. In addition, an initial study of caregivers of patients receiving allogeneic-HSCT were able to benefit from a brief, cognitive behavioral stress management treatment approach. A study examining distress in phase I oncology clinical trial patient caregivers highlighted the need for more support for this significantly distressed population. Furthermore, initial results of the qualitative development study for Pep-Pal yielded support for a mobilized platform delivery of resources for caregivers to manage distress because they acknowledged many barriers to engaging in in-person treatment to manage distress.

ELIGIBILITY:
Inclusion Criteria:

1. Women and men ≥ 18 years of age of any ethnicity
2. Must endorse a moderate level of anxiety (e.g. Score above an 8 on the Hospital and Anxiety Depression Scale (HADS))
3. Speak and read in English
4. Caregiver of a patient with auto HSCT who are moving forward with bone marrow transplant or have receive a bone marrow transplant
5. Caregiver of a patient in a Phase I Clinical Trial
6. Caregiver of a patient diagnosed with advanced cancer (stage III or stage IV)
7. No Cognitive or psychiatric conditions prohibiting participation
8. Must meet criteria for being a primary caregiver, defined as, the person in the patient's life who is primarily responsible for care decisions, emotionally invested in the patient's care, provides instrumental care such as transportation for a patient receiving auto-HSCT, enrolled in a phase I oncology clinical trial, or of a patient diagnosed with advanced cancer (stage IV, solid tumor).
9. Have a computer, smartphone, or tablet with internet access

Exclusion Criteria:

1. Caregivers below the age of 18
2. Score below an 8 on the Hospital and Anxiety Depression Scale (HADS)
3. Cannot speak and read in English
4. Patient does not receive a bone marrow transplant
5. Patient is not enrolled in a Phase I clinical trial
6. Patient is not diagnosed with Stage III or Stage IV cancer
7. Cognitive conditions prohibiting participation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
Evaluation of Exit Interviews | 12 weeks
  Qualitative feedback will be gathered from the first 15 Pep-Pal completer's for individual interviews (5 from Phase I group, 5 from Hematopoietic stem cell transplantation (HSCT) group, 5 from medical oncology) upon completion of the follow-up assessments at 12 weeks about usage, acceptability of content, and impressions of using Pep-Pal.
Pep-Pal Self-Report sessions at 12 Weeks | 12 weeks
  The Investigators will assess feasibility by examining recruitment, retention, as well as reasons for refusal, frequency of sessions watched and length of time spent watching each session. Self report usage of peppal: Usage of Pep-Pal will be quantitatively assessed by asking each participant in the intervention group about their usage including frequency; how many times they watched each session and length of viewing for each session (partial or complete). They will be asked to rate level of usage based on a Likert-scale ranging from not at all to very often for each session (0-10). They will be asked to rank order the list of sessions from most helpful to least helpful.
Evaluation of Self-Report Caregiver reported outcomes at Baseline | Week 1
  Hospital Anxiety and Depression Scale-Anxiety subscale (HADS-A)
Evaluation of Self-report caregiver reported outcomes at 12 weeks | Week 12
  Hospital Anxiety and Depression Scale-Anxiety subscale (HADS-A)

SECONDARY OUTCOMES:
Evaluation of Self-report caregiver reported outcomes at baseline | Week 1
  Center for Epidemiologic Studies Depression Scale (CESD)
Evaluation of Self-report caregiver reported outcomes at baseline | Week 1
  Perceived Stress Scale (PSS)
Evaluation of Self-report caregiver reported outcomes at baseline | Week 1
  Female Sexual Function Index (FSFI)
Evaluation of Self-report caregiver reported outcomes at baseline | Week 1
  Male Sexual Health Questionnaire(MSHQ)
Evaluation of Self-report caregiver reported outcomes at baseline | Week 1
  Measure of Current Status (MOCS-A)
Evaluation of Self-report caregiver reported outcomes at 12 weeks | Week 12
  Center for Epidemiologic Studies Depression Scale (CESD)
Evaluation of Self-report caregiver reported outcomes at 12 weeks | Week 12
  Perceived Stress Scale (PSS)
Evaluation of Self-report caregiver reported outcomes at 12 weeks | Week 12
  Female Sexual Function Index (FSFI)
Evaluation of Self-report caregiver reported outcomes at 12 weeks | Week 12
  Male Sexual Health Questionnaire(MSHQ)
Evaluation of Self-report caregiver reported outcomes at 12 weeks | Week 12
  Measure of Current Status (MOCS-A)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole R Amoyal-Pensak, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pensak NA, Carr AL, Jones J, Mikulich-Gilbertson SK, Kutner JS, Kilbourn K, Sannes TS, Brewer BB, Kolva E, Joshi T, Laudenslager ML. A pilot study of mobilized intervention to help caregivers of oncology patients manage distress. Psychooncology. 2021 Apr;30(4):520-528. doi: 10.1002/pon.5597. Epub 2020 Dec 2. PMID 33217070
- [Derived] Carr AL, Jones J, Mikulich Gilbertson S, Laudenslager ML, Kutner JS, Kilbourn K, Sannes TS, Brewer BW, Kolva E, Joshi T, Amoyal Pensak N. Impact of a Mobilized Stress Management Program (Pep-Pal) for Caregivers of Oncology Patients: Mixed-Methods Study. JMIR Cancer. 2019 May 3;5(1):e11406. doi: 10.2196/11406. PMID 31066678